CLINICAL TRIAL: NCT03949686
Title: Erector Spinae Plane Block for Congenital Hip Dislocation Surgery: Randomized Controlled Double Blind Study
Brief Title: Erector Spinae Plane Block for Congenital Hip Dislocation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA6
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Congenital Hip Dysplasia
Keywords: Postoperative Analgesia; Ultrasound guided erector spinae plane block
MeSH Terms: conditions — Hip Dislocation, Congenital | interventions — Saline Solution; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline + Placebo (Sham Comparator): Ultrasound guided 0.5 ml/kg saline injection to erector spinae plane
  Interventions: Drug: Saline Solution
- ultrasound guided erector spinae plane block (Active Comparator): Ultrasound guided 0.5 ml/kg % 0.250 bupivacaine injection to erector spinae plane
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Saline Solution — 0.5 ml/kg saline
  Other Names: saline
  Arms: Saline + Placebo
Drug: Bupivacaine — 0.5 ml/kg %0.25 bupivacaine
  Arms: ultrasound guided erector spinae plane block

SUMMARY:
Developmental dysplasia of the hip (DDH) is one of the major disorder of the pediatric population with an incidence of 3 to 5 per 1000 children. Open surgical reduction of congenital hip dislocation (CHD) is typically performed after an ineffective closed reduction or older than 18 months. Multiple femoral or pelvic osteotomies and tenotomies are performed during this surgical treatment and cause severe postoperative pain. The aim of this study was to evaluate the analgesic effect of ultrasound guided erector spinae plane block (ESP) in pediatric patients undergoing CHD surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing hip dislocation surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases
* Incomplete patient forms
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* ASA III-IV

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability Score (FLACC) | Postoperative first 24hour
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Need for rescue analgesic | 2 hour
  Number of patients who required rescue analgesia in postoperative care unit in the first 2 hour
Need for analgesic | 24 hour
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkoundi A, Bentalha A, Kettani SEE, Mosadik A, Koraichi AE. Erector spinae plane block for pediatric hip surgery -a case report. Korean J Anesthesiol. 2019 Feb;72(1):68-71. doi: 10.4097/kja.d.18.00149. Epub 2018 Aug 24. PMID 30139214
- [Background] Tulgar S, Kose HC, Selvi O, Senturk O, Thomas DT, Ermis MN, Ozer Z. Comparison of Ultrasound-Guided Lumbar Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block for Postoperative Analgesia in Hip and Proximal Femur Surgery: A Prospective Randomized Feasibility Study. Anesth Essays Res. 2018 Oct-Dec;12(4):825-831. doi: 10.4103/aer.AER_142_18. PMID 30662115